# UNIVERSITY OF MICHIGAN CONSENT TO BE PART OF A RESEARCH STUDY

#### 1. KEY INFORMATION ABOUT THE RESEARCHERS AND THIS STUDY

**Study title:** Alternating Urine Redox Status of Consecutive Menstrual Cycles [Uro-001]. **Principal Investigator:** Dr. Daniel S. McConnell, PhD, Associate Research Scientist, Department of Epidemiology, University of Michigan School of Public Health.

**Study Sponsor:** Urobiologics LLC and the Small Company Innovation Program of the Michigan Economic Development Corporation.

You are invited to take part in a research study. This form contains information that will help you decide whether to join the study.

Taking part in this research project is voluntary. You do not have to participate and you can stop at any time. Please take time to read this entire form and ask questions before deciding whether to take part in this research project.

## 2. PURPOSE OF THIS STUDY

This is a study of your urine during your menstrual cycles. The Sponsor of this study believes that urine chemistry is different from one period to the next. Your urine may be more "oxidative" (a chemistry term) in one period. In your next period, your urine may be less "oxidative". This study will test your and other participants' urines to see if this is true.

#### 3. WHO CAN PARTICIPATE IN THE STUDY

**3.1 Who can take part in this study?** Women age 18-30 who do not smoke and do not vape. You should have "regular" periods (i.e., cycle is 25 to 35 days). You should be willing to participate for 6 months.

If you are having sex with men, you should be trying to prevent pregnancy. You and/or your partner should use barrier protection. This means diaphragms or condoms or similar. You cannot be using hormones such as birth control pills (OCPs, "the pill") or hormone-based intra-uterine devices (IUDs) during the study.

**3.2 How many people are expected to take part in this study?** Approximately 40.

#### 4. INFORMATION ABOUT STUDY PARTICIPATION

#### **KEY INFORMATION**

We wish to measure the redox potential of urine in two back-to-back menstrual cycles

- Urine is to be collected on 2 successive mid-cycle nights and pooled
- Urine is to be collected on two successive cycles.

- The full study will include three pairs of successive mid-cycle collections.
- **4.1 What will happen to me in this study?** First you will read this form, ask any questions, and agree to participate by signing this form. At that point, we will assign you a subject (participant) number.

We will give you a detailed instruction sheet about collecting and delivering the urine samples. You will read the instructions today and ask any questions, especially if there is something you do not understand. You will also keep a record of when your period started and when you collected the urines on forms we give you. If you do not wish to do this as instructed, your participation will end.

To see if you qualify for the study, we have to ask you questions. We will give you the list of questions. The list will include questions about your periods. We will also ask about your history of pregnancy, what medications you are or might start taking, and some related medical questions. If you do not wish to answer all the questions, your participation will end. If you wish to continue, we will collect the required answers from you and determine if you qualify for the study.

If you do not qualify, your participation will end. However, if it seems likely that your answers would be different later and you still want to participate in this study, we will discuss that possibility with you. You would have to give a new consent at that time.

If you decide to participate, you are volunteering to collect your overnight urine at home. You will do an overnight collection of urine for <u>two</u> different nights near the midpoint of your period (13 to 17 days after the beginning of your period). During each collection, you will use an eyedropper to take some of your urine and put it in a sealable vial. When you have done this for two periods in a row, you will deliver the 2 vials to one of our offices around campus, or you will mail them.

We ask you to notify us when your period starts so that we may send you reminders to collect urine at the midpoint of your cycle. If you wish to receive a reminder, please tell us how you want it (by phone call, text, or email). If you do not want reminders or want us to stop reminding you at any time, let us know. (Our contact info is in Section 9, below.)

When you deliver your urine samples, we make sure the vials are labelled with your subject number. From then on, we do not use your name or any identifying information about you. The urine vials will be labeled with only a barcode. Your personal identification will not be present on the urine vials.

We take some urine from each vial and put it in small tubes. The tubes will be assigned a random number (sort of like flipping a coin). We will send the small tubes to the study sponsor, Urobiologics LLC. There will be no way for the sponsor to know your name or any information about you. The sponsor will report the test results to us. We will do a statistical analysis (without using your name) to see if urine chemistry alternates from cycle to cycle.

Testing your urine for oxidative status is experimental. It is not a standard test like you might have in a doctor's office. Your results are important to our research but will have no value or meaning to you.

**4.2** How much of my time will be needed to take part in this study? Because you are collecting your urines at home, the time involved is small. It may take you a minute to set out the collection cups and vials that we give you. It may take you a few minutes longer than usual whenever you pee overnight to collect your urine in a cup and transfer some with the eyedropper to the sealable vial. It may take you a minute to fill out the form with relevant dates. After you collect urine in two consecutive periods, you will deliver both samples to us. If you work or take classes at the University, you may find our drop-off sites convenient. It could take 5 to 15 minutes to bring your urine to the drop-off site. If you prefer to prepare the specimen for mailing, that could take 5 to 15 minutes.

After the time you spend here today, you are being asked to collect urine overnight twice during each of six periods. We estimate setting up and receiving each of 6 reminders may take as much as five minutes, each of 12 overnight collections may take as much as 10 minutes, and each of 3 deliveries may take as much as 15 minutes. Therefore, your total time for this study is 3 to 4 hours. You may require more or less than that to complete your part of the study.

You will have completed the study when you deliver three pairs of urines in the vials provided. Each pair has to be composed of samples that were obtained in two consecutive periods. You may leave the study at any time. We may cancel your participation in the study early if we receive enough total urine samples, if our testing indicates that the study will not work out or the results of the study will be negative, if you are taking too many months to obtain the required paired collections, or for other reasons.

# 5. INFORMATION ABOUT STUDY RISKS AND BENEFITS

**5.1** What risks will I face by taking part in the study? What will the researchers do to protect me against these risks? Collecting and delivering urine should have no risks beyond those of normal daily life. Therefore, participating in this study has minimal, if any, risk to you.

However, because this study collects information about you, the primary risk of this research is a loss of confidentiality. See Section 8 below in this document for more information on how the study team will protect your confidentiality and privacy.

**5.2** How could I benefit if I take part in this study? How could others benefit? You will not receive any personal benefits from being in this study. At this early stage of research, the results will not have any meaning or clinical benefit to you and we will not be providing you with your results. However, others may benefit from the knowledge gained from this study. If our study results are positive, future studies may provide further

knowledge about menstrual cycles and possibly fertility. In any case, we thank you for helping us with this research.

## 6. ENDING THE STUDY

# 6.1 If I want to stop participating in the study, what should I do?

You are free to leave the study at any time. If you leave the study before it is finished, there will be no penalty to you. You will not lose any benefits to which you may otherwise be entitled. If you decide to leave the study before it is finished, please let us know (see Section 9 "Contact Information", below). If you choose to tell us why you are leaving the study, your reasons may be kept as part of the study record. We will keep the information and urine collected from you for the research unless you ask us to remove the information from our records and destroy the urine. If we have already used your information in a research analysis, it will not be possible to remove your information.

## 7. FINANCIAL INFORMATION

- **7.1 Will I be paid or given anything for taking part in this study?** You will receive up to \$125 for your participation in the study as follows: For pairs of urine samples that you obtain as instructed and deliver to us, you will receive \$25 for the first pair, \$50 for the second pair, and \$50 for the third pair. If you leave the study before completing it, you will be paid depending on how many pairs we receive. You will receive MasterCard gift cards. If you prefer a check at the end of your participation in the study, please tell us.
- **7.1.1 Will I need to pay anything to be part of the study?** There should be no cost to you to participate. If you decide to pay for parking to deliver the samples, we will not reimburse it. (We offer a free mail-in option.)
- **7.2 Who could profit or financially benefit from the study results?** As with most research studies, the investigator and research personnel will be paid for their time and effort, and there are costs for equipment and miscellaneous items. These costs are being paid jointly by Urobiologics LLC and the Small Company Innovation Program of the Michigan Economic Development Corporation. The outcome of this study has no effect on the costs and payments. No one on the University research team has any financial interest in the sponsor or in the study outcome.

The study was designed jointly by the sponsor and the University research team. If the study outcome is positive, the sponsor expects to profit from the use of the laboratory method in future. The University and its research team will not profit or get any direct benefit regardless of the study outcome.

Research can lead to new discoveries, such as new tests, drugs, or devices. You will not have rights to these discoveries or any proceeds from them.

# 8. PROTECTING AND SHARING RESEARCH INFORMATION AND URINE

- **8.1 How will the researchers protect my information?** Any papers with your name or other information that might identify you will be kept in a secure and locked cabinet in a secure University laboratory in a University building with security measures in place. Other papers and urine vials will be labelled with your subject number and cannot be identified as yours except by refering to the secured information. Connecting your personal information to specimens or data is done only as described in this Section 8.
- **8.2 Who will have access to my research records?** There are reasons why information about you may be used or seen by the researchers or others during or after this study. Examples include:
  - University, government officials, study sponsors or funders, auditors, and/or the Institutional Review Board (IRB) may need the information to make sure that the study is done in a safe and proper manner.
  - If you receive \$100 or more for taking part in this study, the University of Michigan
    accounting department may need your name, address, Social Security number,
    payment amount, and related information for tax reporting purposes. (If you receive
    over \$600 from the University in any calendar year, the amount you receive will be
    reported to the IRS.)
- **8.3 What will happen to the information and urine collected in this study?** Your name and other information that can directly identify you will be stored securely and separately. All the research information we collected from you (like the questions we ask at the beginning of the study) and the urine analysis data will be managed and analyzed separately, without using your name or other identifying information (called "de-identified" data).

If the study results are negative, we will destroy your personal information and all other information and urine samples per University guidelines. If the study results are positive, we will keep your personal information (stored securely and separately) until we have published the study and only for as long thereafter as required by the publishing journal. We will keep the de-identified information and urine we collected from you during the study, including information from analyzing your urine, in case it is needed to verify our results or for further research. When the principal investigator determines it is appropriate to do so, we will destroy your personal information and all other information and urine samples per University guidelines.

The results of this study could be published in an article or presentation, but will not include any information that would let others know who you are.

**8.4 Will my information and urine be used for future research or shared with others?** No. Any urine remaining after aliquoting and shipping 10 mL to Urobiologics, will be held at the CLASS lab until the end of the study. Samples are held in a locked and secure cabinet at room temperature. At the end of the study any materials remaining will be destroyed per normal practice, any residual urine will be emptied into the city waste disposal system and the emptied containers will be disposed of as biological waste.

**8.4.1 Public information.** We expect this trial to be registered and may report results on the www.clinicaltrials.gov website. This site will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### 9. CONTACT INFORMATION

Whom can I contact about this study? Please contact the researcher listed below to:

- Obtain more information about the study
- Ask a question about the study procedures
- Report an illness, injury, or other problem (you may also need to tell your regular doctors)
- Leave the study before it is finished
- Express a concern about the study

Principal Investigator: Daniel S. McConnell, PhD

Email: danmcc@umich.edu Phone: 734-763-2461

Study Coordinator: Charles Ellis, MD

Email: cellis@umich.edu Phone: 734-665-0493

If you have questions about your rights as a research participant, or wish to obtain information, ask questions, or discuss any concerns about this study with someone other than the researchers, please contact the following:

University of Michigan Health Sciences and Behavioral Sciences Institutional Review Board (IRB-HSBS)

2800 Plymouth Road, Building 520, Room 1169

Ann Arbor, MI 48109-2800

Telephone: 734-936-0933 or toll free (866) 936-0933 Fax: 734-936-1852

E-mail: irbhsbs@umich.edu

#### **10. YOUR CONSENT**

### **Consent to Participate in the Research Study**

By signing this document, you are agreeing to be in this study. Make sure you understand what the study is about before you sign. We will give you a copy of this document for your records and we will keep a copy with the study records. If you have any questions about the study after you sign this document, you can contact the study team using the information in Section 9 provided above.

I understand what the study is about and my questions so far have been answered. I agree to take part in this study.

| Print Legal Name: | |
|-------------------------------|---|
| Signature: | _ |
| Date of Signature (mm/dd/yy): | |

Please be sure to take your copy of this form with you.